CLINICAL TRIAL: NCT04002921
Title: Evaluation of an Arterial Calcification Score as a Predictive Factor of Anastomotic Leakage in Right Colectomy
Acronym: RIGHTCOLOCALCI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD 086-19
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Right Colectomy
Keywords: right colectomy; calcification; anastomotic leakage
MeSH Terms: conditions — Calcinosis; Anastomotic Leak

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Right colectomy: Patient with scheduled right colectomy and with a documented preoperative scan.

SUMMARY:
Anastomotic leakage is the major postoperative complication in right colectomy. Evaluation of calcification on coeliac trunk and mesenteric arteries on the preoperative CT scan could allow the identification of patient at-risk of postoperative complications.

A monocentric retrospective study performed at CHD Vendée concluded than a calcification score over or equal to 3 was associated with a higher risk of developping an anastomotic leakage.

The aim of this prospective multicentric study is to validate a calcification score based on preoperative CT scan analysis and focussing at coeliac trunk and mesenteric arteries.This study will involve patients operated on with a scheduled right colectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Scheduled right colectomy with restoration of digestive continuity
* Patient who has had or will have a preoperative abdominal-pelvic CT scan with or without contrast injection
* Patient with the ability to understand the protocol and agree to participate in the study.
* Affiliated with a social security system

Exclusion Criteria:

* Patient requiring a right colectomy or ileocaecal resection for chronic inflammatory bowel disease or on long-term corticosteroid therapy
* Patient with a history of colic resection
* Patient under guardianship, curatorship, or deprived of liberty
* Pregnant, postpartum or breastfeeding women
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted for right colectomy in one of the 6 hospitals or clinics.
Sampling Method: Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Total calcification score associated with the occurrence of anastomotic leakage | 6 weeks after surgery
  Sum of the calcification scores of the following 4 segments (≥3) associated with the occurrence of anastomotic leakage within 6 weeks postoperatively.
  4 segments:
  * Ostium of celiac artery
  * Ostium of superior mesenteric artery
  * first segment of superior mesenteric artery
  * distal segment of superior mesenteric artery Each segment will be assigned a score between 0 and 2. Total score range : 0-8

SECONDARY OUTCOMES:
Calcification score of each segment associated with the occurrence of anastomotic leakage | 6 weeks after surgery
  4 segments:
  * Ostium of celiac artery
  * Ostium of superior mesenteric artery
  * first segment of superior mesenteric artery
  * distal segment of superior mesenteric artery Each segment will be assigned a score between 0 and 2.
Morbidities defined according to Clavien-Dindo classification | 6 weeks after surgery
  Morbidities defined according to Clavien-Dindo classification occurring at 6 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, Principal Investigator — CHD Vendée
Locations (12):
- France (12):
  - CHU Angers, Angers
  - Hopital privé de Sévigné, Cesson-Sévigné
  - CH de Challans, Challans
  - CH de Cholet 1 rue Marengo, Cholet
  - Centre Hospitalier de Fougères, Fougères
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Mans
  - Clinique Mutualiste de la Porte de l'Orient, Lorient
  - CHU de Nantes, Nantes
  - Centre Hospitalier de Saint Brieuc, Saint-Brieuc
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Hospitalier Bretagne Atlantique, Vannes